CLINICAL TRIAL: NCT04197765
Title: Accelerated Continuous Theta-burst Stimulation (acTBS) for Suicidal Ideation in the Psychiatric Inpatient Setting: A Pilot Study
Brief Title: acTBS Treatment for Inpatient Subjects With Suicidality
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Andrew F. Leuchter, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-001320
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Suicidality
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Sham (Sham Comparator): All parameters will be programmed in the same way as active treatment, however, the treatment will be delivered on the side of the coil that has an internal (hidden) metal shield that will prevent magnetic energy from reaching the skull and brain. Neither the technician, treating physician, nor the patient, will know whether the treatment was delivered from the sham or active side of the coil. The same auditory and tactile cues will be present during active and sham treatment as electrodes will be placed on the scalps of each participant (whether receiving active or sham treatment) that deliver some electrical sensation.
  Interventions: Device: Sham Comparator
- Active acTBS (Active Comparator): For the first three treatments, the study psychiatrist will set treatment intensity to 90% MT, and gradually increase intensity to 120% MT over 20 seconds to maximize tolerability. Subsequent treatment sessions (treatment 4 and onward) will begin, and remain, at 120% MT.
  Treatment will occur 4-5 times a day, separated by an at least 45-min interval between sessions on consecutive weekdays.
  Interventions: Device: accelerated Thetaburst stimulation

INTERVENTIONS:
Device: accelerated Thetaburst stimulation — We will administer 20-30 treatment sessions over the course of the study. The study technician will place the coil over the Fp2 electrode of a 10-20 International EEG system hair net, to approximate stimulation of the R-OFC). For the first three treatments, the study psychiatrist will set treatment intensity to 90% MT, and gradually increase intensity to 120% MT over 20 seconds to maximize tolerability. Subsequent treatment sessions (treatment 4 and onward) will begin, and remain, at 120% MT.
  Treatment will occur 4-5 times a day, separated by an at least 45-min interval between sessions on consecutive weekdays. We estimate all study-related treatments will be complete in 5-6 weekdays.
  Arms: Active acTBS
Device: Sham Comparator — All parameters will be programmed in the same way as active treatment, however, the treatment will be delivered on the side of the coil that has an internal (hidden) metal shield that will prevent magnetic energy from reaching the skull and brain. Neither the technician, treating physician, nor the patient, will know whether the treatment was delivered from the sham or active side of the coil. The same auditory and tactile cues will be present during active and sham treatment as electrodes will be placed on the scalps of each participant (whether receiving active or sham treatment) that deliver some electrical sensation.
  Arms: Sham

SUMMARY:
This is a pilot study to analyze the benefit of accelerated continuous Transcranial magnetic stimulation for inpatient subjects suffering with suicidal ideation. This study will enroll 40 inpatient subjects recruited from the Resnick Neuropsychiatric hospital. Subjects will be blinded and randomized to active or sham TMS treatment and will receive up to 5 assigned treatments per day. Subjects will also be asked to complete mood surveys throughout their participation. Participation in this study will last 7-10 days depending on scheduling.

DETAILED DESCRIPTION:
1.0 SPECIFIC AIMS

Suicide is a leading cause of death worldwide. In the United States, someone commits suicide every 13 minutes. Few treatments exist apart from in-patient hospitalization, medication, and psychotherapy. Repetitive transcranial magnetic stimulation (rTMS) is an efficacious treatment for major depressive disorder (MDD), and may hold therapeutic potential for suicidality, specifically. Novel treatment methods including accelerated theta-burst stimulation (aTBS) allow compressed treatment times and courses, making aTBS ideally suited to an inpatient environment.

In the accelerated continuous theta-burst stimulation for suicidal inpatients (ACT-SI) pilot study, our objective is to examine the feasibility and therapeutic benefit of adding accelerated cTBS to the right orbitofrontal cortex (R-OFC) to standard inpatient treatment in a proof-of-concept, open-label feasibility study. The hypothesis for this study is that active acTBS will be well-tolerated, and lead to a decrease in suicidal ideation over four treatment days.

2.0 RATIONALE

Suicide is a leading cause of death worldwide. Completed suicide significantly, and negatively, affects the individual's family unit, community, and society. Research examining risk factors suggest access to lethal means, accompanied by a specific intent and plan remain significant indicators of acute risk, while a history of suicidal and parasuicidal behaviors, mental health diagnosis (in particular depression), male gender, and history of abuse are common static risk indicators. Psychiatric and legal interventions, including inpatient admission, typically focuses on limiting access to lethal means, and blunting the effect of life stressors, to the greatest extent possible.

Acutely suicidal patients may remain involuntarily on an inpatient unit to receive psychiatric treatment. Nonetheless, little is known about the best methods to treat suicidality. Clinicians may combine psychotherapy with medication to treat depressive and other underlying psychiatric disorders, but treatment can be lengthy, often obviating full treatment courses in the inpatient setting. Acceptable, efficacious, and efficient interventions, suited to brief inpatient stays are sorely needed.

Repetitive transcranial magnetic stimulation (rTMS) is one form of non-invasive brain stimulation (NIBS) that has demonstrated efficacy in the treatment of depression and some evidence of efficacy for suicidality. FDA approved treatment for major depressive disorder (MDD) typically involves a single session of high frequency (10 Hz) stimulation delivered to the left dorsolateral prefrontal cortex (L-DLPFC), lasting 37.5 min a day over several weeks. Research suggests that longer treatment courses may be associated with improved response, remission, and time to relapse. More recently, the FDA approved theta-burst stimulation (TBS), a novel approach requiring 1-3 minutes of treatment per day. Evidence suggests TBS and conventional high-frequency treatment are equivalent in efficacy5. TBS could therefore abbreviate treatment time, enhancing the capacity of an overburdened healthcare system.

Some investigators have also examined the efficacy of rTMS and TBS delivered in an "accelerated" fashion. In this approach a patient receives several sessions (ranging from 2-5) a day with the aim of compressing overall treatment length. Preliminary evidence suggests accelerated TBS (aTBS) may improve suicidal ideation4,8,9 apart from its antidepressive effects8.

TBS is arguably uniquely suited to acceleration, as briefer stimulation sessions allow additional sessions per day, without significantly increasing burden of care. TBS may also have a more favourable safety profile than conventional rTMS10. Moreover, TBS studies in the motor cortex demonstrate a more robust post-stimulation effect on cortical excitability than conventional rTMS. Whether these effects translate into greater therapeutic gains, however, remains undetermined. It was shown that accelerated intermittent TBS (aiTBS) produced an antisuicidal effect in medication-free, treatment resistant depressed outpatients. In their study, there was no separation from sham control, however, the study sample was small, and lack of statistical power along with a high placebo response rate could account for the lack difference observed.

Although most accelerated protocols target the L-DLPFC using excitatory stimulation (i.e. high-frequency, or intermittent theta-burst stimulation [iTBS]), some literature suggests inhibitory rTMS (1 Hz) delivered to the right orbitofrontal cortex (R-OFC) can improve depressive symptoms in those who failed to respond to standard rTMS approaches. Continuous TBS (cTBS) is known to have inhibitory properties15 but unlike standard 1 Hz protocols, can be delivered in under 1 minute. Given its inhibitory properties, and brief administration time, it may be possible to increase stimulation intensity beyond 120% motor threshold, potentially enhancing therapeutic effect, without decreasing tolerability.

To date, the has not been a study that has examined the feasibility and clinical effects of daily R-OFC accelerated cTBS (acTBS) on suicidal ideation in the inpatient setting. This is a proof-of-concept, randomised, sham-controlled pilot study to examine the feasibility (recruitment, retention, tolerability) and clinical effects of acTBS on suicidal thinking in adults admitted to the inpatient unit for suicidality.

3.0 METHODOLOGY

Study Design. The aims to recruit and randomize 40 inpatients (18-65y) with "suicidality" as a reason for admission at the Resnick Neuropsychiatric Hospital to receive: a) active acTBS of the R-OFC or b) sham acTBS of the R-OFC as an add-on intervention to standard inpatient treatment.

Study Specific Endpoints.

Subjects will be involuntarily withdrawn if they experience worsening depression, defined as an increase in IDS-Self Report from baseline of more than 25% during two consecutive assessments, or worsening active suicidal intent, defined as an increase in Suicidal Ideation Attributes Scale of 25% or more over two consecutive assessments, or attempted suicide. In addition, missing more than 10% of treatment sessions consecutively (i.e. 2 sessions in a row) or 20% (i.e. 4 sessions) over the study period will also result in study discontinuation. Subjects will also be withdrawn if they are not compliant with study-specific requirements or if they experience a TMS-induced seizure.

Recruitment. Uo to 40 subjects will be recruited from the psychiatric inpatient unit at the Resnick Neuropsychiatric Hospital. Inpatient psychiatrists will refer patients with MDD and suicidality for a 1-hour consultation with Neuromodulation division staff to determine eligibility. If suitable, staff will offer patients an opportunity to participate, and initiate the consent process.

The inpatient team treating the potential study participant will initiate the recruitment process, however, they will not obtain consent. Treating team members may provide potential Subjects with a study brochure to provide them more information. They may identify potential research subjects and obtain verbal permission from these potential subjects for a member of the research team to approach them. Research team members will contact potential subjects interested in hearing more about the study to initiate the informed consent process.

Research team members will offer all eligible inpatients the option to participate. Participation will be voluntary, and based on informed, capable consent. The decision to participate will not affect an inpatients' receipt of treatment or clinical services at the Resnick Neuropsychiatric Hospital. Research team members will inform subjects that they may terminate their participation at any time, without consequence.

Randomization. Subjects will be assigned to a group (sham versus active) randomly by a computer-generated, block-permutation scheme managed by a study team member not directly involved in study assessments or treatment. This person will inform the study technician of a unique participant code that, when entered into the Magventure stimulator using its research interface, will direct the technician to use one side or another of the coil - thereby determining whether the patient receives sham or active treatment - without the technician knowing which side corresponds to which treatment arm.

Blinding. Only the study team member responsible for randomization will know each participant's group assignment (sham versus active) for the duration of the trial. Subjects, psychiatrists and technicians delivering acTBS will not know which treatment subjects receive. At the end of all treatments, the study team will ask subjects if they believe they received active or sham treatment. The study team members will also write down whether they believe study subjects received sham or active treatment.

Motor Threshold (MT).

On the first day of stimulation, the study psychiatrist will explain the process of motor threshold determination, provide a single test pulse to the patient's forearm to demonstrate the sensation of TMS, and proceed to determine each patient's unique motor threshold using single-pulse TMS. Starting with the magnetic coil tangential to the scalp, at 45 degrees to the midsagittal line, the psychiatrist will deliver suprathreshold single pulses to the motor cortical area corresponding to the abductor polllicis brevis (APB) to initiate visible thumb deflections. The MT is the percentage of stimulator output necessary to cause a thumb deflection in 5 out of 10 trials. This process typically takes approximately 10-15 min and serves to titrate stimulation intensity for the whole of the treatment course.

Stimulation Procedure.

The Magventure Therapy System will be used to administer treatment. The Magventure Therapy System (Model r30) is FDA-approved for Major Depressive Disorder and peripheral stimulation. Subjects will receive up to five sessions of acTBS daily, on consecutive weekdays. Subjects will be escorted from the inpatient unit to the TMS suite where a technician will greet them, and set up the stimulation sessions. Subjects will sit comfortably in a semi-reclined chair for the duration of each session. A Magpro X100 will be used for all study-related TMS procedures, coupled with a CoolB60 A/P treatment coil which allows administrators to deliver both active and sham treatment depending on the orientation of the coil.

Sham stimulation mimics both the auditory (a clicking noise) and somatosensory experiences (i.e. tingling sensation on scalp through electrodes that deliver suprathreshold stimulation with each TMS train) associated with receiving active TMS. Prior research suggests that treatment-naïve subjects (and at times study personnel who have received true TMS in the past) are unable to distinguish sham from active TMS using this arrangement.

Accelerated Continuous Theta-Burst Stimulation (acTBS). Between 20-30 treatment sessions will be administered over the course of the study. The study technician will place the coil over the Fp2 electrode of a 10-20 International EEG system hair net, to approximate stimulation of the R-OFC). For the first three treatments, the study psychiatrist will set treatment intensity to 90% MT, and gradually increase intensity to 120% MT over 20 seconds to maximize tolerability. Subsequent treatment sessions (treatment 4 and onward) will begin, and remain, at 120% MT.

Treatment will occur 4-5 times a day, separated by an at least 45-min interval between sessions on consecutive weekdays. It is estimated that all study-related treatments will be complete in 5-6 weekdays.

Justification for acTBS versus the standard of care for MDD

Though standard rTMS treatment consists of daily sessions of 75 cycles of 4 seconds of 10Hz stimulation followed by 26 seconds of rest over 4-6 weeks, this approach is impractical for typical lengths of stay of 5-10 days. By contrast, our experimental acTBS approach will enable us to compress 20-30 treatments into 4-6 days, enabling inpatients to receive a full course of rTMS add-on therapy without lengthening conventional inpatient stays. Accelerated protocols documented in the literature are well-tolerated.

This experimental approach will differ from published accelerated approaches in that it will use acTBS rather than high-frequency or iTBS treatment. This choice could theoretically enhance tolerability and safety as acTBS is generally thought to be inhibitory in nature, as opposed to both high-frequency and iTBS paradigms. Should this approach prove beneficial in mitigating symptoms of suicidal ideation as indexed by the SIDAS, it may result in the identification of a tolerable, and efficacious augmentation strategy to standard inpatient care.

Potential Side Effects. During the consent process, the study psychiatrist will review common side effects and potential adverse events associated with receiving single-pulse and repetitive-TMS.

Subjects who receive TMS using the Magventure Therapy System are subject to the same risks as FDA-approved Clinical TMS treatment. Generally, TMS is considered safe and well-tolerated. However, it can cause some side effects. They may include headaches, scalp discomfort at the site of stimulation, tingling, spasms or twitching of facial muscles or lightheadedness. Unlike electroconvulsive therapy (ECT), TMS is unassociated with any cognitive impairment. On the contrary, people receiving TMS generally demonstrate improved clarity of thought and memory on post-stimulation cognitive tests. Serious side effects are rare and may include seizures, mania particularly in people with bipolar disorder or hearing loss if there is inadequate ear protection during treatment.

Subjects who receive single pulse TMS using our research or clinical device may experience discomfort from the individual or paired pulses and/or a minor muscle twitch during the pulse. There is no risk of seizure with single pulse TMS.

Risks. Individuals studied in this project will be, by definition, experiencing suicidal thoughts and/or have acted on these thoughts prior to admission In the event that the study team grows concerned about worsening suicidal ideation (as defined in study endpoints), the inpatient treatment team will be notified and study participation terminated.

Subjects may experience psychological discomfort by completing questionnaires about their mental health and suicidal ideation.

Participation in this research may also expose patients to potential breaches in confidentiality and privacy. Every effort will be utilized to guard patient information within the limits of the law. By assigning a research ID that is assigned to study-related data, the code to which will be kept in a locked cabinet, in a locked office, to which only study personnel have access.

The primary risk of this treatment protocol is the potential for lack of clinical improvement. Subjects may suffer some fluctuation or worsening of symptoms during treatment. As a safety precaution, participant's symptoms will be monitored during their treatment.

Seizure Risks:

Generalized seizures have been reported with the use of rTMS in the clinical trial literature. The estimated risk of seizure under ordinary clinical use is approximately 1 in 30,000 treatments (0.003% of treatments) or 1 in 1000 patients (0.001% of patients).

Suicide Individuals with the conditions being studied in this project will, by definition, be at risk for suicidal thoughts or actions. In the event that they tell the research staff that they are thinking about killing themselves or answer 'yes' to a question about having thoughts of suicide, the investigator will ask them additional questions about these thoughts. Depending on how intense these thoughts are or how much they feel like harming themselves or others, the research staff may contact their inpatient physician to discuss these thoughts of self-harm. The investigator will proceed with the Suicide protocol by also reporting to the IRB and all other necessary entities.

Benefits Individual. Individuals participating in the study will receive all acTBS treatments gratis, and may experience improved mood and suicidality as a result.

Society. The results obtained may identify a more efficient and effective TMS treatment for MDD, particularly for those hospitalized for suicidal ideation and actions.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients admitted for "suicidality" with a documented diagnosis of MDD
2. Between the ages of 18 and 65
3. No safety concerns endorsed on the Screening 13-item Questionnaire for rTMS Candidates16
4. Have not received single-pulse or repetitive-TMS in the past, i.e. considered "TMS naïve".

Exclusion Criteria:

* (1) lifetime diagnosis of schizophrenia, schizoaffective disorder, delusional disorder, current psychotic symptoms (2) a history of epilepsy or any other major neurological disorder (3) Any exclusion on the 13-item Questionnaire for rTMS Candidates (4) diagnosis of borderline personality disorder, assessed on a case by case basis (5) concomitant major unstable medical illness (6) current withdrawal from psychoactive substances (7) history of failed brain stimulation (i.e. rTMS, ECT, VNS, DBS, TNS in the past)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Suicidal Ideation Attributes Scales (SI-DAS) | Baseline to Final visit
  This 5-item questionnaire is a self-report measure that asks completers to rate the frequency, controllability, closeness to attempt, distress, and interference of suicidal thinking with daily activities from 0-10, with 10 indicating extreme intensity. The SIDAS takes approximately 30-60 seconds to complete and has excellent internal reliability, sensitivity, and specificity. The score is calculated as the sum of the five items. Scores of 21 or above denote high suicidal ideation. A lower score indicates improvement in suicidality.
Change in Inventory of Depressive Symptom (Self-report) | Baseline to final visit
  The 30-item questionnaire used to assess the severity of depressive symptoms. The scale covers symptoms such as as mood reactivity, distinct mood quality, diurnal mood variation, irritable mood, anxious mood, capacity for pleasure, sexual interest, bodily aches and pains, panic or phobic symptoms, digestive problems, interpersonal rejection sensitivity, and leaden paralysis. The sum of the 30 items yields the overall score. A higher score indicates worsening in depressive symptoms. Score ranges from 0 to 84.

CONTACTS AND LOCATIONS:
Locations (1):
- Resnick Neuropsychiatric Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No